CLINICAL TRIAL: NCT03598374
Title: Effects of Oral Inositol Supplementation on Spontaneous Reproductive Outcomes in Infertile Polycystic Ovarian Syndrome Women.
Brief Title: Spontaneous Reproductive Outcomes After Oral Inositol Supplementation in Infertile Polycystic Ovarian Syndrome Women.
Acronym: IROP-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IROP-1
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Polycystic Ovarian Syndrome; Infertility, Female
Keywords: Inositol; Polycystic ovarian syndrome; Fertility; Clinical pregnancy rate; Miscarriage rate; Live birth rate
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female | interventions — Inositol; Folic Acid

STUDY DESIGN:
Intervention Model Description: Randomized multi centre double-blind controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, care provides, investigators and outcome assessors are blinded for the treatment: Inositol + Folic acid versus Folic acid alone. The treatment allocation is identified by code number before the study start, and will be revealed only after data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inositol + Folic acid (Experimental): Couples with PCOS infertile women, diagnosed according to the Rotterdam criteria, who access infertility center with conception desire. These women will receive oral supplementation with Inositol (Myo-inositol and D-chiro-inositol at 40:1 ratio) plus Folic acid for 6 months.
  Couples are required to have regular intercourse with the aim to achieve a spontaneous conception.
  Interventions: Dietary Supplement: Inositol + Folic acid; Behavioral: Regular intercourses
- Folic acid (Placebo Comparator): Couples with PCOS infertile women, diagnosed according to the Rotterdam criteria, who access infertility center with conception desire. These women will receive oral supplementation with Folic acid for 6 months.
  Couples are required to have regular intercourse with the aim to achieve a spontaneous conception.
  Interventions: Dietary Supplement: Folic acid; Behavioral: Regular intercourses

INTERVENTIONS:
Dietary Supplement: Inositol + Folic acid — Daily oral supplementation of for 6 months or until pregnancy conception:
  Myo-Inositol: 1100 mg D-chiro-inositol: 27.6 mg Folic acid: 400 mcg
  Arms: Inositol + Folic acid
Dietary Supplement: Folic acid — Daily oral supplementation of for 6 months:
  Folic acid: 400 mcg
  Arms: Folic acid
Behavioral: Regular intercourses — Couples are required to have regular intercourses with the aim to achieve a spontaneous conception.

SUMMARY:
Polycystic ovarian syndrome (PCOS) is a heterogeneous, multifaceted and complex disorder characterized by insulin resistance (IR), hyperinsulinemia, and hyperandrogenism leading ovarian disfunction and infertility. Given the central pathogenic role of IR in the endocrine, reproductive, and metabolic disturbances of PCOS, several pharmacological and non-pharmacological approaches have been proposed to counteract the hyper insulinemic IR typical of the syndrome. Two Inositol stereoisomers, Myo-Inositol (MI) and D-chiro-inositol (DCI), captured the attention of researchers for their insulin-sensitizing actions, which configure them as proper candidates for the treatment of PCOS.

Very few studies reported on spontaneous clinical pregnancy rates, none were powered for this outcome, and none reported on the clinically relevant outcome of live birth. Therefore, data about clinical pregnancy rate, live birth rate, and miscarriage rate comparing inositols with placebo are limited.

Conversely, about infertility and assisted reproduction techniques (ART), improvements have been reported in PCOS women who underwent fertility treatment using inositol in different forms, combinations or doses. This data, considering the different tissue-specific ratios (i.e., 100:1 in the ovary) and the different physiological roles of inositol stereoisomers, suggest that DCI supplementation alone might not be the optimal or appropriate approach for improving IVF outcomes in PCOS patients, and drawn attention to the importance of MI and DCI supplementation in a physiological ratio in order to restore normal ovary functionality. Indeed, the combination of MI and DCI, at a more physiological ratio of 40:1, was able to more quickly restore to normal the hormonal and metabolic parameters in PCOS women than MI treatment alone or DCI treatment alone, improving the endocrine profile and IR of women with PCOS.

Nevertheless, regarding infertility the primary outcomes that should be considered are clinical pregnancy rate, miscarriage rate and live birth rate. Although many studies showed improved hormonal and metabolic profile and improved ovulation rate and higher quality and number of oocyte retrieved in ART in PCOS women after inositols administration, data about clinical pregnancy rate, live birth rate, and miscarriage rate are limited with several concerns regarding interpretation of the studies.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS diagnosed by Rotterdam criteria in couple that desire to conceive.

Exclusion Criteria:

* Male infertility factor that require in vitro fertilization technique.
* Women with infertility factors that require in vitro fertilization technique.
* Couple with infertility factors that require in vitro fertilization technique.
* Diabetes mellitus that require insulin or oral drugs treatment.
* Any other pre-pregnancy or pregnancy-induced/related disease.
* Any other pharmacological, non-pharmacological or nutraceutical treatment (beside oral folic acid supplementation) more than 3 months before the enrollment (wash-out period) or during the trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Within 6 months from the enrollment
  Number of spontaneous pregnancies conceived per women diagnosed by transvaginal ultrasound. Diagnosis is based on the identification of intrauterine gestational sac with embryo and/or yolk sac.
Miscarriage rate | Within 6 months from the enrollment
  Number of spontaneous abortion per women diagnosed by positive pregnancy test with subsequent spontaneous interruption of the pregnancy.
Live birth rate | Within 18 months from the enrollment
  Number of spontaneous pregnancies per women resulted in a delivered viable fetus.
Spontaneous ovulation rate | Change in spontaneous ovulation rate, through study completion (an average of 18 months)
  Spontaneous ovulation activity evaluated by menstrual cycle regularization. Menstrual cycles evaluated by intervals between menstruations (days), day of menstrual blood flow. Rate evaluate considering the number of women with restored regular menstrual cycles per women with irregular menstrual cycles.

SECONDARY OUTCOMES:
Glucose metabolism | Change in glucose metabolism, through study completion (an average of 18 months)
  OGTT: values of oral glucose tolerance test. Impaired glucose metabolism is diagnosed if fasting glucose values were abnormal (100-125 mg/dl) or glucose tolerance is impaired (2 h plasma glucose within OGTT range of 140-199 mg/dl), and when glucose values exceed threshold values for gestational diabetes (fasting glu- cose value ≥92mg/dl, 1-hour glucose value ≥180mg/dl or 2- hour glucose value ≥153mg/dl)
BMI | Change in BMI, through study completion (an average of 18 months)
  Body mass index
Lipid metabolism | Change in Lipid metabolism, through study completion (an average of 18 months)
  Lipid profile assessed by evaluation the high density lipoprotein level and triglycerides level.
Blood pressure | Change in Blood pressure, through study completion (an average of 18 months)
  systolic and diastolic blood pressure
Androgens profile | Change in Androgens profile, through study completion (an average of 18 months)
  Serum free testosterone, dehydroepiandrosterone sulfate, and serum SHBG serum concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Simone Garzon, M.D., Principal Investigator — Universita di Verona; Fabio Ghezzi, M.D., Study Chair — Università degli Studi dell'Insubria; Massimo Franchi, M.D., Study Chair — Universita di Verona

IPD SHARING:
Plan to Share IPD: Undecided